CLINICAL TRIAL: NCT03824912
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd) to Ketoconazole Cream 2% (G&W Laboratories Inc.) in the Treatment of Tinea Pedis
Brief Title: Clinical Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% in the Treatment of Tinea Pedis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Encube Ethicals Pvt. Ltd. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry); ACM Global Laboratories (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71875502
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, three-arm, parallel group, multiple-site bioequivalence study with clinical endpoints.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study products are blinded and provided to the patients in the same packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test: Ketoconazole Cream 2% (Experimental): Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)
  Interventions: Drug: Ketoconazole Cream 2%
- Reference: Ketoconazole Cream 2% (Active Comparator): Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)
  Interventions: Drug: Ketoconazole Cream 2% (G&W Laboratories Inc.)
- Placebo: Cream (Test vehicle) (Placebo Comparator): Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketoconazole Cream 2% — Patients will be instructed to apply sufficient study product to cover affected and immediate surrounding areas once daily for 42 ± 4 days. Each patient is expected to receive 42 ± 4 doses.
  Arms: Test: Ketoconazole Cream 2%
Drug: Ketoconazole Cream 2% (G&W Laboratories Inc.) — Patients will be instructed to apply sufficient study product to cover affected and immediate surrounding areas once daily for 42 ± 4 days. Each patient is expected to receive 42 ± 4 doses.
  Arms: Reference: Ketoconazole Cream 2%
Drug: Placebo — Patients will be instructed to apply sufficient study product to cover affected and immediate surrounding areas once daily for 42 ± 4 days. Each patient is expected to receive 42 ± 4 doses.
  Arms: Placebo: Cream (Test vehicle)

SUMMARY:
Clinical Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% in the Treatment of Tinea Pedis

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd) to Ketoconazole Cream 2% (G&W Laboratories Inc.) in the Treatment of Tinea Pedis

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant, non-lactating female, ≥ 18 years of age.
2. Signed informed consent form (ICF) that meets all criteria of current Food and Drug Administration regulations.
3. Female patient of childbearing potential must not be pregnant or lactating at Visit 1 (as confirmed by a negative urine pregnancy test with a sensitivity of less than 50 milli-International unit (mIU/mL) or equivalent units of human chorionic gonadotropin).
4. Female patient of childbearing potential must agree to the use of a reliable method of contraception throughout the study (e.g., total abstinence, intrauterine device, a double-barrier method, oral, transdermal, injected, or implanted non-hormonal or hormonal contraceptive) throughout the study. A sterile sexual partner is not considered an adequate form of birth control. If the female is using any estrogen or oral contraceptive therapy, the same product must have been taken for at least one month before Visit 1.
5. Have clinical diagnosis of tinea pedis with lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot (the non-interdigital lesions should not be hyperkeratotic, i.e., characteristic of tinea pedis moccasin).
6. The presence of tinea pedis infection provisionally confirmed at baseline by a positive potassium hydroxide (KOH) wet mount preparation (i.e., skin scrapings from the target site are placed on a microscope slide with a drop of 10% KOH, and microscopic examination reveals segmented fungal hyphae).
7. The sum of clinical signs and symptoms scores of the target lesion ≥ 4. See Appendix A for scoring scale:

   1. Signs: Fissuring/cracking, erythema, maceration and scaling
   2. Symptoms: pruritus and burning/stinging In addition the target lesion must have a minimum score ≥ 2 for erythema and a minimum score ≥ 2 for either pruritus or scaling.

Exclusion Criteria:

1. Females who are pregnant, lactating or planning to become pregnant during the study period.
2. History of or current psoriasis, Lichen planus or contact dermatitis involving the feet within the previous 12 months.
3. History of dermatophyte infections with a lack of response to antifungal therapy (recurrent tinea pedis [i.e., more than 3 infections in the past 12 months] that were unresponsive to previous antifungal therapy).
4. History of allergy, hypersensitivity, or intolerance to ketoconazole, other imidazoles, sulfites or any other component of the study product.
5. Confluent, diffuse moccasin-type tinea pedis of the entire plantar surface.
6. Current uncontrolled diabetes.
7. Presence of any other infection of the foot or other disease process that, in the Investigator's opinion, may interfere with the evaluation of the patient's tinea pedis.
8. Known history of or current impaired wound healing, presence of peripheral vascular disease and/or trophic changes of the lower limbs to an extent that, in the opinion of the Investigator, would make the patient unsuitable for the study or compromise patient's safety.
9. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder, immunosuppression (due to disease or therapy, including history of organ transplant), or other medical condition that, in the Investigator's opinion, would place the patient at undue risk by participating or compromise the integrity of the study data.
10. Use of antipruritics, including antihistamines, within 72 hours before Visit 1.
11. Use of topical corticosteroids, topical antibiotics or topical antifungal therapy (e.g., clotrimazole, econazole, fluconazole) within 2 weeks before Visit 1.
12. Use of systemic (e.g., oral or injectable) antibiotics, systemic antifungal therapy, or systemic corticosteroids within 30 days before Visit 1. The use of intranasal, inhaled or ophthalmic corticosteroids for acute or chronic conditions (e.g., allergic conjunctivitis, asthma/chronic obstructive pulmonary disease maintenance) is acceptable to the extent that, in the opinion of the Investigator, does not compromise safety of patient or integrity of data.
13. Use of oral terbinafine or itraconazole within 2 months before Visit 1.
14. Use of immunosuppressive medication or radiation therapy within 3 months before Visit 1.
15. Receipt of any drug as part of a research study within 30 days before Visit 1.
16. Previous participation in this study.
17. Employee of the Investigator or research center or their immediate family members.
18. Inability to understand the requirements of the study and the relative information or are unable or unwilling to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lalatendu Panigrahi, Study Director — Encube Ethicals Pvt. Ltd.
Locations (9):
- United States (7):
  - Long Beach Clinical Trial Services, Inc., Long Beach, California
  - International Dermatology Research, Inc., Miami, Florida
  - FXM Research Corp., Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - FXM Research Miramar, Miramar, Florida
  - MOORE Clinical Research, Inc., Tampa, Florida
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania
- FXM Research International, Belize City, Belize
- FXM Research International, Castries, Saint Lucia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2% | Placebo: Cream (Test Vehicle)
Started | 332 | 335 | 164
Completed | 192 | 201 | 96
Not Completed | 140 | 134 | 68
Not completed — Lost to Follow-up | 18 | 15 | 8
Not completed — Negative Baseline Culture Result | 118 | 112 | 57
Not completed — Non-Compliance with Study Drug | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 4 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Participation in another study | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population was used for the baseline analysis population. The Safety population included all randomized patients who used at least one dose of product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2% | Placebo: Cream (Test Vehicle) | Total
Number analyzed (Participants) | 314 | 319 | 156 | 789
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (13.6) | 46.7 (13.9) | 44.8 (14.4) | 45.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 114 | 64 | 309
  Male | 183 | 205 | 92 | 480
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 154 | 153 | 75 | 382
  Not Hispanic or Latino | 160 | 166 | 81 | 407
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 147 | 153 | 74 | 374
  White | 166 | 163 | 80 | 409
  More than one race | 1 | 3 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: The Number of Patients in Each Treatment Group With a Therapeutic Cure of Tinea Pedis (Equivalence: Per-Protocol Population)
Description: Equivalence: Per-Protocol Population Therapeutic Cure: To be considered a Therapeutic Cure, the patient must have both Clinical and Mycological Cure of tinea pedis.
  Therapeutic Failure: A patient will be considered a Therapeutic Failure if:
  1. the patient is a Clinical or Mycological Failure
  2. the patient was considered to have an insufficient therapeutic response
  3. the patient used topical drug therapy for irritation or pruritus on the feet after the treatment phase of the study
Time Frame: Two weeks after the end of treatment (Day 56 ± 4) (Equivalence)
Population: The Per-Protocol population was used for this analysis to determine equivalence between the Test and Reference groups only. To determine equivalence, only the test and reference treatment arms are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2%
Number analyzed (Participants) | 184 | 191
Participants | 89 | 90

2. Primary Outcome: Primary Efficacy Endpoint: The Number of Patients in Each Treatment Group With a Therapeutic Cure of Tinea Pedis (Superiority: Modified Intent-to-Treat Population)
Description: Superiority: modified Intent-to-Treat Population Therapeutic Cure: To be considered a Therapeutic Cure, the patient must have both Clinical and Mycological Cure of tinea pedis.
  Therapeutic Failure: A patient will be considered a Therapeutic Failure if:
  1. the patient is a Clinical or Mycological Failure
  2. the patient was considered to have an insufficient therapeutic response
  3. the patient used topical drug therapy for irritation or pruritus on the feet after the treatment phase of the study
Time Frame: Two weeks after the end of treatment (Day 56 ± 4) (Superiority)
Population: The MITT Population was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2% | Placebo: Cream (Test Vehicle)
Number analyzed (Participants) | 195 | 199 | 97
Participants | 92 | 94 | 26

3. Secondary Outcome: Secondary Efficacy Endpoint: The Number of Patients in Each Treatment Group With a Clinical Cure of Tinea Pedis (Equivalence: Per-Protocol Population)
Description: Clinical Cure: To be considered a clinical cure the patient's total severity score must be ≤ 2 with no individual severity score > 1.
  Clinical Failure: A patient will be considered a Clinical Failure if the patient's total severity score is > 2 or any individual score is > 1.
  Local Signs and Symptoms The most severely affected area will be identified as the target lesion at the baseline visit and will be used for the assessments at Day 42 and Day 56 visits.
  The Clinical Signs and Symptoms of tinea pedis will be rated by the Investigator as "none", "mild," "moderate" or "severe" using the following standardized rating scale.
  0 = None (complete absence of any sign or symptom)
  1. = Mild (Slight)
  2. = Moderate (Definitely Present)
  3. = Severe (Marked, Intense)
  The following signs and symptoms will be rated at each visit:
  * Signs: Fissuring/cracking, erythema, maceration, and scaling
  * Symptoms: Pruritus and burning/stinging
Time Frame: Two weeks after the end of treatment (Day 56 ± 4) (Equivalence)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2%
Number analyzed (Participants) | 184 | 191
Participants | 97 | 110

4. Secondary Outcome: Secondary Efficacy Endpoint:The Number of Patients in Each Treatment Group With a Mycological Cure of Tinea Pedis (Equivalence: Per-Protocol Population)
Description: Mycological Cure: To be considered a mycological cure the patient must have a negative Potassium hydroxide (KOH) test and a negative fungal culture.
  Mycological Failure: A patient will be considered a Mycological Failure if the patient's KOH test is positive or the patient's fungal culture is positive.
Time Frame: Two weeks after the end of treatment (Day 56 ± 4) (Equivalence)
Population: The PP population was used for this analysis to determine equivalence between the Test and Reference groups only. One patient had an inconclusive result for the fungal culture at Visit 3 and was excluded from the analysis of the secondary endpoint for the mycological cure. Patient was a clinical failure and was included in the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2%
Number analyzed (Participants) | 184 | 190
Participants | 127 | 118

5. Secondary Outcome: Secondary Efficacy Endpoint: The Number of Patients in Each Treatment Group With a Clinical Cure of Tinea Pedis (Superiority: Modified Intent-to-Treat Population)
Description: as for outcome 3
Time Frame: Two weeks after the end of treatment (Day 56 ± 4) (Superiority)
Population: The MITT population was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2% | Placebo: Cream (Test Vehicle)
Number analyzed (Participants) | 195 | 199 | 97
Participants | 100 | 116 | 35

6. Secondary Outcome: Secondary Efficacy Endpoint:The Number of Patients in Each Treatment Group With a Mycological Cure of Tinea Pedis (Superiority: Modified Intent-to-Treat Population)
Description: as for outcome 4
Time Frame: Two weeks after the end of treatment (Day 56 ± 4) (Superiority)
Population: The MITT population was used for the analysis. One patient had an inconclusive result for the fungal culture at Visit 3 and was excluded from the analysis of the secondary endpoint for the mycological cure. Patient was a clinical failure and was included in the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2% | Placebo: Cream (Test Vehicle)
Number analyzed (Participants) | 195 | 198 | 97
Participants | 132 | 122 | 39

ADVERSE EVENTS:
Time Frame: 5 months
Description: The "Total Number of Participants at Risk" is not consistent with the numbers provided in any of the rows in the Participant Flow module, since the Overall Summary of Adverse Events is based on the Safety Population.
  The Safety population will include all randomized patients who use at least one dose of product.
Arm/Group | Test: Ketoconazole Cream 2% | Reference: Ketoconazole Cream 2% | Placebo: Cream (Test Vehicle)
All-Cause Mortality (participants affected / at risk) | 0/314 | 0/319 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/314 | 0/319 | 0/156
Other Adverse Events (participants affected / at risk) | 12/314 | 15/319 | 6/156
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test: Ketoconazole Cream 2% (N=314) | Reference: Ketoconazole Cream 2% (N=319) | Placebo: Cream (Test Vehicle) (N=156)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 5 (6) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the Clinical Trials Agreements between the sites and the Contract Research Organization, sites are instructed that the Investigator shall not publish, or seek to publish, either in whole or in part any results of the Study without the written consent.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT03824912/SAP_000.pdf
  • Study Protocol (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT03824912/Prot_001.pdf